CLINICAL TRIAL: NCT06659861
Title: An Exploratory Randomized Comparative Study to Evaluate the Effect of RV3278B-OS0386 on Skin Ecosystem, in Teenagers with Mild to Moderate Facial Acne
Brief Title: Efficacy of Cosmetic Product RV3278B-OS0386 on Skin Surface Ecosystem, in Teenagers with Mild to Moderate Facial Acne
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pierre Fabre Dermo Cosmetique (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RV3278B20240316
Record Dates: First submitted 2024-10-21; First posted 2024-10-26 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Acne
Keywords: Skin ecosystem; cosmetic care product
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test Group (Experimental): This group will apply the RV3278B-OS0386 cosmetic product for acne prone skin.
  Interventions: Other: RV3278B-OS0386
- Control Group (Other): This group will receive the associated cosmetic product RV4632A-RY1845 (emollient cream), to be applied in the event of facial skin discomfort only.
  Interventions: Other: RV4632A-RY1845

INTERVENTIONS:
Other: RV3278B-OS0386 — Cosmetic product to be applied twice a day on the face during the whole study
  Arms: Test Group
Other: RV4632A-RY1845 — Cosmetic product to be applied in the event of facial skin discomfort only
  Arms: Control Group

SUMMARY:
The aim of this exploratory study is to better understand the mechanisms of action of the RV3278B-OS0386 cosmetic product on the cutaneous ecosystem, in acne context.

DETAILED DESCRIPTION:
This study will be conducted as an exploratory monocentric, randomized, comparative study.

A total number of 52 subjects (teenagers with mild to moderate facial acne) will be included and randomized in two parallel groups :

* The tested group who will apply the tested product RV3278B-OS0386
* The control group who will not apply the tested product. However, they will receive the associated product (RV4632A-RY1845), to be applied in the event of facial skin discomfort only.

  3 visits are planned:
  * Visit 1 (Day 1) : Inclusion, randomization, collection of biological samples on the forehead and start of product application.
  * Visit 2 (Day 29 +/- 3 days) : Phone call follow-up
  * Visit 3 (Day 57, a window of + 3 days is allowed): End-of-study visit - Collection of biological samples on the forehead.

ELIGIBILITY:
Inclusion Criteria:

Criteria related to the population:

* Female and male aged between 12 and 17 years included
* Subject having signed his/her written informed consent/assent for his/her participation in the study
* Subject whose parent(s) or guardian(s) has (have) given his/her (their) written consent for their child's participation in the study
* Subject affiliated to a social security system or health insurance, or is a beneficiary
* Subject whose parent(s) or guardian(s) is (are) registered with health social security or health insurance
* Subject and/or parents certifying the truth of the personal information declared to the investigator
* Cooperative subject and/or parent(s)/legal representative(s), aware of the necessity and duration of controls so that perfect adhesion to the protocol established by the clinical trial centre could be expected
* Subject with phototype I, II, III, IV according to the Fitzpatrick scale
* For woman/girl of childbearing potential:

  * use of an effective method of contraception, as assessed by the investigator, introduced and unchanged for at least 1 month (3 months in case of hormonal contraception) before inclusion in the study
  * accept to go on using it during the whole duration of the study

Criteria related to the skin condition (acne):

* Subject with combination, combination to greasy skin tendency or oily skin on face
* Subject with mild to moderate acne vulgaris on face; GEA from 2 to 3
* Subject with predominantly non-inflammatory acne on the forehead
* Subject with at least 20 open comedones on the face, excluding the nose area, at the inclusion

Subject presenting on his/her forehead (extension possible to the temples, but excluding the hair): target areas suitable for study samplings and measurements:

Inclusion criteria required for at least 26 subjects:

• Subject having a sensitive skin, according to his/her own self-assessment

Criteria related to the treatments and/or products:

• Subject who used the same facial cleansing product, shaving products, make-up (if applicable) for at least 1 month before inclusion and is willing to keep it during the whole duration of the study

Non Inclusion Criteria:

Criteria related to the population:

* Subject unable to understand the information given including study procedures (for linguistic or psychiatric reasons) and to give his/her consent in writing and to report required information in writing in his/her diary
* Subject whose parent(s) or guardian(s) is(are) unable to understand the information given (for linguistic or psychiatric reasons) and to give his/her consent in writing
* For woman of childbearing potential: pregnant or breastfeeding or planning to be pregnant during the study
* Subject who has forfeited his/her freedom by administrative or legal award or is under guardianship
* Subject whose parent(s) or guardian(s) who has forfeited his/her freedom by administrative or legal decision or under guardianship
* Subject or parent(s)/legal representative(s) not able to be contacted in case of emergency
* Subject who, in the judgement of the investigator, is not likely to be compliant with study-related constraints and requirements
* Subject whose parent(s) or guardian(s) is(are) unable to comply with study-related constraints
* Subject admitted in a sanitary or social facility
* Subject planning an hospitalization during the study
* Subject who is currently participating, who plans to participate or who has participated within the previous weeks or months in another clinical study liable to interfere with the study assessments according to the investigator's assessment
* Subject is in a position likely to represent a conflict of interest and/or is a family member of any people involved in the conduct of the study (secretary, nurse, technician,…), of the investigational site

Criteria related to the subject's health / skin condition:

* Subject with history of allergy or intolerance to any of the study products ingredients
* Subject with history of allergy or intolerance to any material used for the research (like pen, pencil, marker pen, sticking plaster…)
* Subject having any other dermatologic condition than acne, or characteristics (like tattoo) on the study area(s) liable to interfere with the study assessments
* Subject having a dermatological condition, an acute, chronic or progressive disease or history of disease liable to interfere with the study data or considered by the Investigator hazardous for the subject or incompatible with the study requirements
* Presence of more than an acne inflammatory nodule in the whole face
* Clinical signs of hormone dysfunction or hyperandrogenism
* Severe form of acne (acne conglobate, acne fulminans or nodulocystic acne) or acneiform eruptions, in the investigator's opinion
* Exposure to UV-Rays or excessive exposure to sunlight within the previous month

Criteria related to treatments and/or products:

* Any surgery, chemical (e.g.: skin peel) or physical treatment on the face in the 12 months before the inclusion visit or planned during the study
* Systemic isotretinoin treatment taken in 6 months before the inclusion or planned during the study
* Systemic acne treatment (e.g., zinc gluconate, antibiotics, hormonal treatment [excluding contraception] …] taken in the 3 months before the inclusion or planned to be taken during the study
* Probiotics taken orally in the month before the inclusion or planned to be taken during the study
* Use of self-tanning product on the face in the month before the inclusion or planned to be used during the study
* Topical acne treatment (e.g., benzoyl peroxide, vitamin A and its derivates) applied on the face in the month before the inclusion or planned during the study
* Topical or systemic Non-Steroidal Anti-Inflammatory (NSAI), corticosteroids, taken or applied to the face in the 2 weeks before the inclusion or planned to be taken/applied during the study
* Change in subject's usual make-up, facial hygiene habits, cleansing products, care products, shaving products and/or use new products on the face in the 2 weeks before the inclusion visit or planned during the study
* Skincare product for acne (e.g., product containing any ingredient, like "anti-blemish" active ingredient, liable to interfere with the study according to investigator's assessment) applied to the face in the 2 weeks before the inclusion visit or planned to be applied during the study
* Home care on the face (including exfoliation, masks, home peels, etc.) used in the 2 weeks before the inclusion visit or planned to be used during the study
* Any topical or systemic treatment established or modified during the previous weeks or planned to be established or modified during the study, liable to interfere with the assessments performed during the study according to the investigator's opinion
* Last face shaving performed in the 2 days before the inclusion visit
* Any topical treatment or product (including make-up) applied to the face between the last wash (performed the day before the visit) and the inclusion visit
* Water applied on the face within 8 hours before the inclusion

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-03-06 (Actual); Study Completion 2025-03-06 (Actual)

PRIMARY OUTCOMES:
Effect of the RV3278B on acne severity | Change from Visit 1 (Day 1) to Visit 3 (Day 57).
  Assessed by the investigator on a 6-point scale (0 to 5 with 0: clear and 5: very severe)
Effect of the RV3278B on open comedones. | Change from Visit 1 (Day 1) to Visit 3 (Day 57).
  Quantification of open comedones
Effect of the RV3278B on biological criteria within isolated comedones | Change from Visit 1 (Day 1) to Visit 3 (Day 57).
  Analyses of comedone composition
Effect of the RV3278B on biological criteria from the skin surface | Change from Visit 1 (Day 1) to Visit 3 (Day 57).
  Analyses of skin microbiota
Effect of the RV3278B on biometrological criteria | Change from Visit 1 (Day 1) to Visit 3 (Day 57).
  Skin potential hydrogen measurement by pH meter
Adverse events related to RV3278B | From Visit 1 (Day 1) to Visit 3 (Day 57)
  Adverse events occurrence will be determined by the subject's/parent(s) or guardian(s) spontaneous reporting, the investigator's non-leading questioning and his/her clinical evaluation

SECONDARY OUTCOMES:
Illustrative Outcome : Standardized photographs of the subject's face | Visit 1 (Day 1) to Visit 3 (Day 57).

CONTACTS AND LOCATIONS:
Locations (1):
- Cidp Romania, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: No